CLINICAL TRIAL: NCT03741621
Title: Viscosity Rather Than Quality of Dietary Fibre Predicts Cholesterol-lowering Effect in Healthy Individuals
Brief Title: Viscosity of Fibre Predicts Cholesterol-lowering in Healthy Individuals
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Kellogg Company (Industry); University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: viscosity and cholesterol
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Lipidemia; Healthy
Keywords: dietary fibre; Viscosity; lipids; Healthy
MeSH Terms: conditions — Hyperlipidemias | interventions — Psyllium; Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Viscosity (Experimental): viscous fibre blend added to breakfast cereals consumed in the context of a typical North American diet for 3 weeks duration
  Interventions: Dietary Supplement: Viscous Fibre Blend
- Medium Viscosity (Experimental): Kellogg's Bran buds with psyllium breakfast cereal consumed in the context of a typical North American diet for 3 weeks duration
  Interventions: Dietary Supplement: Psyllium
- Low Viscosity (Experimental): Kellogg's All Bran breakfast cereal consumed in the context of a typical North American diet for 3 weeks duration
  Interventions: Dietary Supplement: Wheat Bran

INTERVENTIONS:
Dietary Supplement: Viscous Fibre Blend — High viscosity viscous fiber blend sprinkled on wheat and maize bran cereals(Bran Buds®; Kellogg Company)
  Arms: High Viscosity
Dietary Supplement: Psyllium — Bran Buds cereal (white bran and maize bran) with psyllium (Bran Buds® with PSY; Kellogg Company)
  Arms: Medium Viscosity
Dietary Supplement: Wheat Bran — All Bran cereal (All Bran®; Kellogg Company)
  Arms: Low Viscosity

SUMMARY:
To investigate the role of fibre viscosity (low, medium, high) in lowering cholesterol in healthy individuals

ELIGIBILITY:
Inclusion Criteria:

-healthy individuals

Exclusion Criteria:

* regular alcohol consumption
* regular smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 1992-01 (Actual); Primary Completion 1994-01 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
change in LDL cholesterol | change from baseline after 21 days, relative to control

SECONDARY OUTCOMES:
change in total cholesterol | change from baseline after 21 days, relative to control
change in triglycerides | change from baseline after 21 days, relative to control
change in HDL cholesterol | change from baseline after 21 days, relative to control
change in apolipoprotein B | change from baseline after 21 days, relative to control
change in apolipoprotein A-1 | change from baseline after 21 days, relative to control